CLINICAL TRIAL: NCT06816875
Title: Comparative Analysis of Commercially Available Nasal Aspirators in Infants
Brief Title: Comparison of the User Experience of Four Nasal Aspirators in Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Dr. Noze Best LLC (Unknown)
Responsible Party: Principal Investigator, Valerie Cote, Physician, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHEO REB# 25/07X
Record Dates: First submitted 2025-01-27; First posted 2025-02-10 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Upper Respiratory Tract Infection
Keywords: nasal aspirator in infants; user experience of nasal aspirators
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- NozeBot Arm (Experimental): Participants assigned to this group will receive the NozeBot electric nasal aspirator device.
  Interventions: Device: NozeBot Electric Nasal Aspirator
- NoseFrida Arm (Active Comparator): Participants assigned to this group will receive NoseFrida the SnotSucker product.
  Interventions: Device: NoseFrida the SnotSucker
- hydraSense Arm (Active Comparator): Participants assigned to this group will receive the hydraSense Baby Nasal Aspirator Starter Kit.
  Interventions: Device: hydraSense Baby Nasal Care Nasal Aspirator Starter Kit
- Braun Arm (Active Comparator): Participants assigned to this group will receive the Braun nasal aspirator device.
  Interventions: Device: Braun Nasal Aspirator

INTERVENTIONS:
Device: NozeBot Electric Nasal Aspirator — The NozeBot is a rechargeable, battery-operated baby nasal aspirator with a nosepiece that loops directly onto the caregivers fingers for ease of use, and is intended to be held so it sits just inside the nose to create a seal. It will be used according to its manufacturer's instructions for use in this study.
  Arms: NozeBot Arm
Device: NoseFrida the SnotSucker — The NoseFrida is nose-to-mouth nasal suctioning device with a disposable hygienic filter. The nosepiece is a larger tube that is to be held so it sits against and not inside the nose to create a seal. It will be used according to its manufacturer's instructions for use in this study.
  Arms: NoseFrida Arm
Device: hydraSense Baby Nasal Care Nasal Aspirator Starter Kit — The hydraSense Baby Nasal Aspirator Starter Kit is a nose-to-mouth nasal suctioning device with a disposable hygienic filter. The kit contains pre-proportioned saline solution vials to liquify mucus prior to suctioning. The nosepiece is intended to be held so it sits inside the nose to create a seal. It will be used according to its manufacturer's instructions for use in this study.
  Arms: hydraSense Arm
Device: Braun Nasal Aspirator — The Braun nasal aspirator is a battery-operated nasal suctioning device with a washable collection chamber for mucus. There are two nosepiece sizes to accommodate a best fit in the nose. It will be used according to its manufacturer's instructions for use in this study.
  Arms: Braun Arm

SUMMARY:
The goal of this clinical trial is to compare the caregiver's user experience, and overall impacts on an infant's cold symptoms between four nasal aspirator devices. These devices are normally used to relieve congestion in infants. when they are sick by softening and suctioning mucus from the nose.

The main questions it aims to answer are:

What is the caregiver's user experience of the NozeBot electric nasal aspirator compared to three commonly accessible nasal aspirator devices?

Are there changes in the infant's sleeping, feeding, or breathing as reported by the caregiver when using the NozeBot compared to the three other nasal aspirator devices?

Are there changes in their caregiver's habits when using the NozeBot compared to the three other nasal aspirator devices?

Researchers will compare the self-reported measures of caregiver's user experience, reported changes to their infant's symptoms, and reported changes to their own sleeping and care habits between the NozeBot electric nasal aspirator and three comparator devices: the NoseFrida SnotSucker, the hydraSense Baby Nasal Aspirator Kit, and the Braun electric nasal aspirator.

Participants will be assigned to receive one of the four devices at the start of their participation. They will be asked to use the assigned device at home according to the device instructions during two periods: (1) for 10 days while their infant is sick, and (2) for up to 3 months after.

During these periods, participants will be asked to complete online surveys at predetermined intervals to report the user experience, any changes to their infant's sleeping, feeding or breathing, and any changes to their own sleeping habits and perceived stress levels. These intervals for survey completion are: (i) after 1-2 days of use while their infant is sick, (ii) after 4-5 days of use while their infant is sick, (iii) after 7-10 days of use while their infant is sick, and then (iv) biweekly for 3 months.

ELIGIBILITY:
Inclusion Criteria

A parent(s)/caregiver(s)/family will be eligible to participate if:

* They have a child between 2 months - 18 months of age
* They are seeking outpatient care for that child for a respiratory illness (cold, flu, RSV) at the Kids Come First Care clinic
* The child does not have any contraindications to the use of a nasal aspirator
* The parent(s)/caregiver(s) are fluent in English

Exclusion Criteria

A parent(s)/caregiver(s)/family will be ineligible to participate if:

* They have a child younger than 2 months or 13 months old or older currently seeking outpatient care for a respiratory illness
* The child is admitted to hospital
* The child does not have a respiratory illness
* The child has a diagnosed craniofacial syndrome
* The child has a defined contraindication and cannot use a nasal aspirator
* The parents/caregivers are not comfortable using a nasal aspirator
* The parent/caregivers are not fluent in English

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Differences in the caregiver's user experience on device ease of use between the NozeBot and the NoseFrida, hydraSense and Braun devices | This is reported at all follow ups, from the first survey completed at 1-2 days of device use to the final survey completed at the end of the third month of use per participant
  The first measure of user experience is the self-reported rating by the caregivers on the ease of use of the device, including device set up, use, and cleaning after use. This is reported on a 5-point Likert scale (1 - difficult to 5 - easy) at each of the survey follow ups.
Differences in the caregiver's satisfaction between the NozeBot and the NoseFrida, hydraSense and Braun devices | This is reported at the 7-10 days of device use to the final survey completed at the end of the third month of use per participant.
  The second measure of user experience is the caregiver-reported satisfaction with the device, including confidence that the device is helping their infant, and that the device's power is sufficiently removing mucus. This is reported on a 5-point Likert scale (1 - very dissatisfied to 5 - very satisfied) once at the 7-10 days of use while their child is sick, and at each bi-weekly survey over the 3 months.
Differences in the caregiver's reported net promoter score between the NozeBot and the NoseFrida, hydraSense and Braun devices | This is reported at the 7-10 days of device use to the final survey completed at the end of the third month of use per participant.
  The third measure of user experience is the a rating by the caregiver on whether they would recommend the device to someone when their child is sick (also known as Net Promoter Score). This is reported on a 5-point Likert scale (1 - very unlikely to 5 - very likely) once at the 7-10 days of use while their chlid is sick, and at each bi-weekly survey over the 3 months.

SECONDARY OUTCOMES:
Self-reported changes in the caregiver's sleep habits between the NozeBot and the NoseFrida, hydraSense and Braun devices | This is reported at the 1-2 days of use, 4-5 days of use, and 7-10 days of use follow up surveys.
  Recorded as self-reported perceived changes to the caregivers' sleeping habits during the time that their child is sick since they started using the device in the study. This is reported on a 5-point Likert scale (1 - much less than normal to 5 - a lot more than normal) at the 1-2 days of use, 4-5 days of use, and 7-10 days of use follow up surveys.
Self-reported changes in the caregiver's perceived ability to care for their sick child between the NozeBot and the NoseFrida, hydraSense and Braun devices | This is reported at all follow ups, from the first survey completed at 1-2 days of device use to the final survey completed at the end of the third month of use per participant
  Recorded as self-reported perceived changes to the caregivers' ability to take care of their child during the time that their child is sick since they started using the device in the study. This is reported on a 5-point Likert scale (1- much less able to 5 - a lot more capable) at each of the survey follow ups.
Self-reported changes in the caregiver's perceived stress levels while caring for a sick child between the NozeBot and the NoseFrida, hydraSense and Braun devices | This is reported at all follow ups, from the first survey completed at 1-2 days of device use to the final survey completed at the end of the third month of use per participant
  Recorded as self-reported perceived changes to the caregivers' stress levels experienced while their child is sick since they started using the device in the study. This is reported on a 5-point Likert scale (1- strongly disagree to 5 - strongly agree) at each of the survey follow ups.
Caregiver-reported changes in their infant's sleeping habits between the NozeBot and the NoseFrida, hydraSense and Braun devices | This is reported at the 1-2 days of use, 4-5 days of use, and 7-10 days of use follow up surveys.
  Reported as caregiver-rated perceived changes in their infant's sleeping habits since they started using the device in the study on a 7-point Likert scale (1 - sleeping much worse to 4 - no changes in sleep to 7 - sleeping much better).
Caregiver-reported changes in their infant's feeding habits between the NozeBot and the NoseFrida, hydraSense and Braun devices | This is reported at the 1-2 days of use, 4-5 days of use, and 7-10 days of use follow up surveys.
  Reported as caregiver-rated perceived changes in their infant's feeding habits since they started using the device in the study on a 7-point Likert scale (1 - much harder to feed to 4 - no changes to feeding to 7 - much easier to feed).
Caregiver-reported perceived changes in their infant's breathing between the NozeBot and the NoseFrida, hydraSense and Braun devices | This is reported at all follow ups, from the first survey completed at 1-2 days of device use to the final survey completed at the end of the third month of use per participant
  Reported as caregiver-rated perceived changes in their infant's breathing since they started using the device in the study on a 4-point Likert scale (1 - no change in breathing to 4 - breathing a lot better).

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this research may be used in future related research projects that are either an extension of the original project or in the same general area of research (secondary use of data). Researchers outside of this specific study may request access to the coded database for new research purposes with a specific study plan and agreement to use the coded data only for that research. Participants will not be asked to provide additional informed consent for the use of their coded data for future research. As this study is being conducted to compare the user experience of the NozeBot to three competitor devices, future data sharing requests will be reviewed and allowed in collaboration with Dr. Noze Best.
Access Criteria: Researchers and research teams with a study plan can request access to the coded IPD and supporting information. An agreement to use the data only in accordance with the study plan will be put in place to allow electronic access.